CLINICAL TRIAL: NCT06698042
Title: A Phase 3 Randomized, Open-label Clinical Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous Pembrolizumab Coformulated With Hyaluronidase (MK-3475A) Versus Intravenous Pembrolizumab, in the First-line Treatment of Participants With Metastatic Non-small Cell Lung Cancer With PD-L1 TPS 50% or Greater
Brief Title: A Clinical Study of Pembrolizumab (+) Berahyaluronidase Alfa (MK-3475A) to Treat Newly-diagnosed Metastatic Non-small Cell Lung Cancer (MK-3475A-F84)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-F84; MK-3475A-F84 (Other: MSD); 2024-513165-39-00 (Registry Identifier: EU CT); U1111-1306-1214 (Registry Identifier: UTN); jRCT2031240445 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (+) Berahyaluronidase alfa (Experimental): Pembrolizumab (+) Berahyaluronidase alfa SC will be administered for squamous and nonsquamous NSCLC as per the schedule specified in arm; participants may be eligible for second course.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa
- Pembrolizumab (Active Comparator): "Pembrolizumab by IV Infusion will be administered for squamous and nonsquamous NSCLC as per the schedule specified in arm; participants may be eligible for second course,
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab (+) Berahyaluronidase alfa — Administered subcutaneously on Day 1 of each cycle
  Other Names: MK-3475A
  Arms: Pembrolizumab (+) Berahyaluronidase alfa
Biological: Pembrolizumab — Administered intravenously on Day 1 of each cycle
  Other Names: MK-3475; KEYTRUDA®; SCH 900475
  Arms: Pembrolizumab

SUMMARY:
Researchers are looking for new ways to treat non-small cell lung cancer (NSCLC) that is metastatic, which means cancer has spread to other parts of the body.

Some people with metastatic NSCLC are treated with pembrolizumab, an immunotherapy treatment that is given into a vein as an intravenous (IV) infusion. Pembrolizumab (+) Berahyaluronidase alfa is pembrolizumab that is given under the skin as a subcutaneous (SC) injection. The goal of this study is to learn what happens to pembrolizumab in a person's body over time when it is given as an IV infusion or SC injection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous or nonsquamous non-small cell lung cancer (NSCLC).
* Measurable disease as assessed by the local site investigator/radiology.

Exclusion Criteria:

* Diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements.
* Received prior systemic anticancer therapy for their metastatic NSCLC.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2030-02-11 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of Pembrolizumab Measured After the First Dose | At designated time points (up to approximately 14 months)
  AUC is defined as area under curve exposure. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine AUC.
Trough Concentration (Ctrough) of Pembrolizumab Measured at Steady State | At designated time points (Up to ~15 months)
  Ctrough is defined as the trough concentration at steady-state. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough

SECONDARY OUTCOMES:
Number of Participants Who Experience an AE- All Participants | Up to approximately 28 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 25 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (67):
- United States (4):
  - Providence Medical Foundation ( Site 0117), Fullerton, California
  - Illinois Cancer Care ( Site 0101), Peoria, Illinois
  - Montefiore Medical Center ( Site 0104), The Bronx, New York
  - University of Cincinnati Medical Center ( Site 0112), Cincinnati, Ohio
- China (18):
  - Beijing Peking Union Medical College Hospital ( Site 5000), Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital ( Site 5018), Chongqing, Chongqing Municipality
  - Fujian Province Cancer Hospital ( Site 5007), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 5008), Xiamen, Fujian
  - The first affiliated hospital, Sun Yat-Sen university ( Site 5011), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 5003), Guangzhou, Guangdong
  - Huizhou Central People's Hospital ( Site 5004), Huizhou, Guangdong
  - Jiangmen Center Hospital ( Site 5001), Jiangmen, Guangdong
  - Liuzhou People's Hospital ( Site 5009), Liuchow, Guangxi
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 5015), Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University ( Site 5019), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital ( Site 5014), Changchun, Jilin
  - Jinan Central Hospital ( Site 5012), Jinan, Shandong
  - Shanghai Pulmonary Hospital ( Site 5010), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 5016), Chengdu, Sichuan
  - Sichuan Cancer Hospital. ( Site 5006), Chengdu, Sichuan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine ( Site 5021), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 5002), Linhai, Zhejiang
- Germany (2):
  - HELIOS Klinikum Erfurt ( Site 2005), Erfurt, Thuringia
  - Universitätsklinikum Jena ( Site 2002), Jena, Thuringia
- Guatemala (4):
  - MEDI-K ( Site 1101), Guatemala City
  - CELAN,S.A ( Site 1104), Guatemala City
  - Private Practice- Dr. Rixci Augusto Lenin Ramírez ( Site 1102), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 1103), Quetzaltenango
- Japan (13):
  - Fujita Health University Hospital ( Site 4004), Toyoake, Aichi-ken
  - Ehime University Hospital ( Site 4007), Tōon, Ehime
  - Hospital of the University of Occupational and Environmental Health, Japan ( Site 4010), Kitakyushu, Fukuoka
  - Takarazuka City Hospital ( Site 4006), Takarazuka, Hyōgo
  - Kanagawa Cardiovascular and Respiratory Center ( Site 4002), Yokohama, Kanagawa
  - Kochi Medical School Hospital ( Site 4012), Nankoku, Kochi
  - Miyagi Cancer Center ( Site 4000), Natori-shi, Miyagi
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 4009), Sakai, Osaka
  - Saitama Prefectural Cancer Center ( Site 4001), Kitaadachi-gun, Saitama
  - Tochigi Cancer Center ( Site 4008), Utsunomiya, Tochigi
  - Juntendo University Hospital ( Site 4003), Bunkyo, Tokyo
  - Fukushima Medical University Hospital ( Site 4011), Fukushima
  - Osaka International Cancer Institute ( Site 4005), Osaka
- Peru (4):
  - Clínica San Antonio ( Site 1006), Trujillo, La Libertad
  - Clínica Internacional - Sede San Borja ( Site 1002), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 1004), Lima
  - Oncosalud ( Site 1000), Lima
- Poland (2):
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 2305), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii ( Site 2303), Warsaw, Masovian Voivodeship
- Romania (4):
  - SC Radiotherapy Center Cluj SRL ( Site 2203), Floreşti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 2201), Craiova, Dolj
  - Spitalul Municipal Schuller Ploiești ( Site 2204), Ploieşti, Prahova
  - Institutul Oncologic ( Site 2202), Cluj-Napoca
- South Korea (3):
  - Pusan National University Hospital ( Site 3002), Pusan Kwangyokshi, Pusan-Kwangyokshi
  - Chungnam National University Hospital ( Site 3003), Daejeon, Taejon-Kwangyokshi
  - Korea University Guro Hospital ( Site 3001), Seoul
- Spain (5):
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 2454), Donostia / San Sebastian, Gipuzkoa
  - Hospital General Universitari Vall d Hebron ( Site 2450), Barcelona
  - INSTITUTO CATALAN DE ONCOLOGIA- L´HOSPITALET DE LLOBREGAT ( Site 2451), Barcelona
  - Hospital Universitario Juan Ramon Jimenez ( Site 2453), Huelva
  - Hospital Universitario Virgen Macarena ( Site 2455), Seville
- Turkey (Türkiye) (6):
  - Ege Universitesi Hastanesi-Chest Diseases Department ( Site 2501), Bornova, İzmir
  - Gulhane Egitim Arastirma Hastanesi ( Site 2504), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2500), Ankara
  - Gazi University Health Research and Application Center Gazi Hospital-Oncology ( Site 2502), Ankara
  - Ankara Bilkent Sehir Hastanesi ( Site 2503), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi ( Site 2506), Istanbul
- United Kingdom (2):
  - Torbay Hospital ( Site 2100), Torquay, England
  - The Royal Cornwall Hospital ( Site 2102), Truro, England

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26348&tenant=MT_MSD_9011